CLINICAL TRIAL: NCT06765980
Title: A Phase 1/2, First-in-Human, Multi-Arm, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Efficacy of an Adeno-associated Virus Vector VV-14295 Administered Suprachoroidally With the Everads Injector In AdultS With GeographIc Atrophy Secondary to Age-related Macular DegeneratiON (the VISION Study)
Brief Title: A Study to Evaluate KRIYA-825 (VV-14295) in Adults With Geographic Atrophy Secondary to Age-related Macular Degeneration
Acronym: VISION
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kriya Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KRIYA-825-101
Record Dates: First submitted 2024-12-19; First posted 2025-01-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: Geographic Atrophy Secondary to Age-related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Part 1a, low dose (Experimental): A single low dose of VV-14295 will be administered on Day 1. In addition, oral prednisone and difluprednate eye drops will be administered prior to and after VV-14295 dosing to reduce the risk of inflammation. After several weeks, participants will switch from difluprednate to prednisolone acetate eye drops.
  Interventions: Genetic: VV-14295
- Part 1a, high dose (Experimental): A single high dose of VV-14295 will be administered on Day 1. In addition, oral prednisone and difluprednate eye drops will be administered prior to and after VV-14295 dosing to reduce the risk of inflammation. After several weeks, participants will switch from difluprednate to prednisolone acetate eye drops.
  Interventions: Genetic: VV-14295
- Part 1b (Experimental): A single dose of VV-14295 determined from Part 1a will be administered on Day 1. In addition, oral prednisone and difluprednate eye drops will be administered prior to and after VV-14295 dosing to reduce the risk of inflammation. After several weeks, participants will switch from difluprednate to prednisolone acetate eye drops.
  Interventions: Genetic: VV-14295
- Part 2 (Experimental): A single dose of VV-14295 determined from Part 1a will be administered on Day 1. In addition, oral prednisone and difluprednate eye drops will be administered prior to and after VV-14295 dosing to reduce the risk of inflammation. After several weeks, participants will switch from difluprednate to prednisolone acetate eye drops.
  Interventions: Genetic: VV-14295

INTERVENTIONS:
Genetic: VV-14295 — VV-14295 will be administered as a single suprachoroidal injection.

SUMMARY:
The goal of this study is to evaluate how safe and tolerable KRIYA-825 (VV-14295) is and to determine how effective it is in reducing the growth of geographic atrophy (GA) lesions in the treated eye in patients with GA secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be between 55 to 80 years of age (inclusive), at the time of signing the informed consent form.
* Body mass index (BMI) of 19 to 34 kg/m2 (inclusive).
* Must agree to use reliable contraception for at least 12 months after administration of VV-14295. A female participant is eligible to participate if she is not pregnant and not breastfeeding.
* The GA lesion must meet certain criteria as assessed by a central reading center's assessment of imaging at Screening.
* Adequate clarity of ocular media, adequate pupillary dilation, and fixation to permit the collection of good quality images as determined by the Investigator.
* For study eye, Normal Luminance BCVA of 55 letters or worse using the ETDRS charts (20/80 or worse) for Part 1a participants or 24 letters or better (approximately 20/320 Snellen equivalent) for Part 1b and Part 2 participants.
* Fellow eye Normal Luminance BCVA of 5 letters or better using ETDRS charts (20/800 or better) for Part 1a participants or 24 letters or better (approximately 20/320 Snellen equivalent or better) for Part 1b and Part 2 participants. Fellow eye must have equivalent or better visual acuity than the study eye.

Exclusion Criteria:

* Any ocular disease or condition that is not GA secondary to AMD: Macular atrophy secondary to a condition other than AMD; Exudative AMD diagnosis or any history of or active macular neovascularization (in study eye or fellow eye) and/or retinal angiomatous proliferation associated with AMD or any other cause; Presence of an active ocular disease that in the opinion of the Investigator compromises or confounds visual function; Active ocular or periocular infection or active uncontrolled intraocular inflammation within 3 months of Screening; History of vitrectomy, retinal detachment, or corneal transplant in the study eye; Active/history of uveitis.
* Any ocular condition that prevents adequate imaging.
* Medical, cognitive or psychiatric conditions that, in the opinion of the Investigator, make consistent study assessment and follow-up over the 12-month Post-Treatment Follow-up Period unlikely, or could increase the risk to the participant by participating in the study or confound the outcome of the study.
* Hospitalization within 1 year prior to Screening that, in the opinion of the Investigator, make consistent study assessment and follow-up over the 12-month Post-Treatment Follow-up Period unlikely, or could increase the risk to the participant by participating in the study or confound the outcome of the study.
* Any Screening test (e.g., ECG) or laboratory value (e.g., hematology) that in the opinion of the Investigator and/or Medical Monitor is clinically significant and renders the participant not suitable for study participation.
* Participant has a direct contraindication to the steroid regimen (both oral and topical) or has a condition that significantly increases the risk of complication.
* Active/history of malignancy within the past 5 years from Screening or any previous therapeutic radiation in the region of the study eye(s) at Screening. History of non-melanoma skin cancers (e.g., basal cell, squamous cell carcinomas), cervical intraepithelial neoplasia (CIN), and localized prostate cancer after treatment are not exclusionary.
* Intraocular surgery (including lens replacement surgery) within 3 months prior to Screening.
* History of laser therapy in the macular region.
* History of intravitreal (IVT) therapy, such as IVT steroid injections, within 6 months prior to Screening.
* COVID-19 vaccine within 90 days of Screening or plan to receive COVID-19 vaccine within 6 months of treatment.
* Active use of systemic immunomodulatory drugs or systemic corticosteroids in the last 60 days. Topical steroids are not exclusionary.
* Prior participation in another interventional clinical study for GA within the past 12 months from the last dosing at Screening.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular and non-ocular adverse events, abnormal clinical laboratory values, abnormal physical examinations, abnormal vital signs, abnormal electrocardiograms (ECGs), and abnormal ophthalmic findings | 12 months
  Evaluate Part 1 safety of VV-14295 in foveal and non-foveal patients
Incidence and severity of ocular and non-ocular adverse events, abnormal clinical laboratory values, abnormal physical examinations, abnormal vital signs, abnormal ECGs, and abnormal ophthalmic findings | 12 months
  Evaluate Part 2 safety of VV-14295 in non-foveal GA patients
Rate of GA progression as assessed by optical coherence tomography (OCT) | 12 months
  Part 2 efficacy of VV-14295

SECONDARY OUTCOMES:
Rate of GA progression as assessed by fundus autofluorescence (FAF) | 3, 6, and 12 months
  Parts 1 and 2 efficacy of VV-14295
Rate of GA progression as assessed by OCT | 3, 6, and 12 months
  Parts 1 and 2 efficacy of VV-14295
Visual function preservation as assessed by best-corrected visual acuity (BCVA) | 3, 6, and 12 months
  Parts 1 and 2 efficacy of VV-14295
Visual function preservation as assessed by low luminance visual acuity (LLVA) | 3, 6, and 12 months
  Parts 1 and 2 efficacy of VV-14295
Visual function preservation as assessed by microperimetry | 3, 6, and 12 months
  Parts 1 and 2 efficacy of VV-14295
VV-14295 transgene product expression | 12 months
  Concentrations of AAV vector-mediated transgene product in serum
Immune response to VV-14295 | 12 months
  Humoral and cellular responses to AAV2 capsid and transgene product; anti-AAV2 neutralization capacity in serum
Vector shedding profile of VV-14295 | 12 months
  Vector shedding in serum, tears, mucus, and urine
Safety of Everads Injector | 1 day post-dose
  Frequency of device-related adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- Kriya Clinical Study Site, Ottawa, Ontario, Canada
- Kriya Clinical Study Site, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No